CLINICAL TRIAL: NCT06135649
Title: A Prospective Lymphadenectomy Protocol to Investigate the Pattern of Nodal Spread and Its Association With Oncologic Outcomes in Post-neoadjuvant Pancreatoduodenectomy
Brief Title: Dissecting the Pattern of Nodal Spread in Post-neoadjuvant Pancreatoduodenectomy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Universita di Verona (Other)
Responsible Party: Principal Investigator, Giuseppe Malleo, Associate Professor of Surgery, Universita di Verona
Other Study IDs: LN_NAT
Record Dates: First submitted 2023-11-12; First posted 2023-11-18 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Pancreas Cancer; Pancreatic Adenocarcinoma
Keywords: Pancreatoduodenectomy; Lymphadenectomy; Lymph nodes; Pancreatic cancer
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Systematic lymphadenectomy — The nodal dissection protocol included the ISGPS lymphadenectomy stations (5, 6, 8a, 12b-c, 13, 14a-b, and 17) extended to stations contiguous to the regional basin (8p, 12a-p, and jejunal mesentery nodes). Stations embedded in the PD specimen (13, 14a-b, 17 and jejunal mesentery LN) were defined as first nodal echelon, while stations sampled as distinct specimens (5, 6, 8a-p, 12a-b-p-c) were defined as second nodal echelon.

SUMMARY:
There has been long-standing debate about nodal dissection in pancreatoduodenectomy (PD) for pancreatic ductal adenocarcinoma (PDAC), with most studies examining the value of nodal yields, number of metastatic nodes and spatial location of metastases being conducted in the upfront surgery setting. With increasing use of a chemotherapy-first approach even in early stage PDAC, the validity of nodal parameters in post-treatment PD has been brought into question due to therapy-induced lymph node (LN) shrinkage. However, the available information is based on retrospective data or administrative registries, which only considered the number of examined and metastatic nodes, without detailed information regarding the dissection protocol and the influence of nodal metastases location. Back in 2013, corresponding to the standard lymphadenectomy definition release by the International Study Group of Pancreatic Surgery (ISGPS) and the diffusion of multi-agent chemotherapy regimens, an institutional, station-based nodal dissection protocol was established for post-neoadjuvant PD. The aim was to investigate whether the pattern of metastatic spread within the nodal basin is a superior quality metric for prognosis relative to the count-based classification system.

ELIGIBILITY:
Inclusion Criteria:

* Post-neoadjuvant pancreatoduodenectomy for localized pancreatic ductal adenocarcinoma.

Exclusion Criteria:

* Oligometastatic disease
* Upfront pancreatectomy
* Incomplete lymphadenectomy
* Macroscopically incomplete resections
* Rare variants of pancreatic cancer

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Consecutive patients with localized pancreatic ductal adenocarcinoma receiving post-neoadjuvant pancreatoduodenectomy from June 2013were eligible for inclusion in the study.
Sampling Method: Non-Probability Sample
Enrollment: 850 (Estimated)
Dates: Start 2013-01 (Actual); Primary Completion 2019-12 (Actual); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Metastatic involvement of second nodal echelon | 3 years
  Rate of metastases to nodes outside the main resection specimen (stations 6,8,12)

SECONDARY OUTCOMES:
Metastatic involvement of single nodal stations | 8 years
  Rate of metastases in each station included in the lymphadenectomy protocol
Overall survival | 3 years
  Overall survival from pancreatectomy stratified by nodal echelon
Recurrence-free survival | 3 years
  Recurrence-free survival from pancreatectomy stratified by nodal echelon
Overall survival | 8 years
  Overall survival from pancreatectomy stratified by nodal stations
Recurrence-free survival | 8 years
  Recurrence-free survival from pancreatectomy stratified by nodal stations

CONTACTS AND LOCATIONS:
Locations (1):
- Unit of Pancreatic Surgery - G.B. Rossi Hospital, University of Verona Hospital Trust, Verona, VR, Italy

IPD SHARING:
Plan to Share IPD: Undecided
Data will be available upon reasonable request.

REFERENCES:
- [Background] Malleo G, Maggino L, Capelli P, Gulino F, Segattini S, Scarpa A, Bassi C, Butturini G, Salvia R. Reappraisal of Nodal Staging and Study of Lymph Node Station Involvement in Pancreaticoduodenectomy with the Standard International Study Group of Pancreatic Surgery Definition of Lymphadenectomy for Cancer. J Am Coll Surg. 2015 Aug;221(2):367-79.e4. doi: 10.1016/j.jamcollsurg.2015.02.019. Epub 2015 Feb 28. PMID 26081176
- [Background] Malleo G, Maggino L, Casciani F, Lionetto G, Nobile S, Lazzarin G, Paiella S, Esposito A, Capelli P, Luchini C, Scarpa A, Bassi C, Salvia R. Importance of Nodal Metastases Location in Pancreatoduodenectomy for Pancreatic Ductal Adenocarcinoma: Results from a Prospective, Lymphadenectomy Protocol. Ann Surg Oncol. 2022 Jun;29(6):3477-3488. doi: 10.1245/s10434-022-11417-3. Epub 2022 Feb 21. PMID 35192154
- [Background] Malleo G, Maggino L, Qadan M, Marchegiani G, Ferrone CR, Paiella S, Luchini C, Mino-Kenudson M, Capelli P, Scarpa A, Lillemoe KD, Bassi C, Castillo CF, Salvia R. Reassessment of the Optimal Number of Examined Lymph Nodes in Pancreatoduodenectomy for Pancreatic Ductal Adenocarcinoma. Ann Surg. 2022 Nov 1;276(5):e518-e526. doi: 10.1097/SLA.0000000000004552. Epub 2020 Nov 9. PMID 33177357
- [Background] Javed AA, Ding D, Baig E, Wright MJ, Teinor JA, Mansoor D, Thompson E, Hruban RH, Narang A, Burns WR 3rd, Burkhart RA, Lafaro K, Weiss MJ, Cameron JL, Wolfgang CL, He J. Accurate Nodal Staging in Pancreatic Cancer in the Era of Neoadjuvant Therapy. World J Surg. 2022 Mar;46(3):667-677. doi: 10.1007/s00268-021-06410-y. Epub 2022 Jan 7. PMID 34994834
- [Background] Arrington AK, O'Grady C, Schaefer K, Khreiss M, Riall TS. Significance of Lymph Node Resection After Neoadjuvant Therapy in Pancreatic, Gastric, and Rectal Cancers. Ann Surg. 2020 Sep 1;272(3):438-446. doi: 10.1097/SLA.0000000000004181. PMID 32740236